CLINICAL TRIAL: NCT05119283
Title: Clinical Study of a Formulation Containing Phtalox® for the Prevention and Control of Periodontal Disease
Brief Title: Clinical Study of a Formulation Containing Phtalox® in Periodontal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Alfenas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Phtalox in Periodontal Disease
Record Dates: First submitted 2021-10-20; First posted 2021-11-15 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Periodontal Diseases; Periodontitis; Bone Loss
Keywords: Oral Antiseptic; Mouth Rinse; Periodontal treatment
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Bone Diseases, Metabolic | interventions — Mouthwashes

STUDY DESIGN:
Intervention Model Description: Thirty patients will be recruited who will undergo scaling and coronal-root planing (RAR), and after basic periodontal treatment will be randomly divided into 3 groups according to the supporting treatment: G1 - patients who will receive mouthwashes with saline solution; G2 - patients who will receive 0.12% chlorhexidine mouthwash; G3 - patients who will be treated with PHTALOX®.
Masking Description: After basic periodontal treatment, patients will be randomly divided based on a draw with closed, opaque and non-translucent envelopes, into 3 groups according to the supporting treatments: G1 - patients who will receive mouthwashes with saline solution; G2 - patients who will be rinsed with 0.12% chlorhexidine and G3 - patients who will be treated with PHTALOX®. Each group will consist of the same number of patients, that is, 10. Patients will receive 140 mL of the substances, to be used for 7 days, twice a day.
  Clinical reassessments of patients will be made before the treatments, and at 15, 30 and 60 after the performance of the RAR and beginning of the respective mouthwashes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phtalox (Experimental): Patients will undergo scaling and coronal-radicular smoothing and rinses with PHTALOX mouthwashes.
  Interventions: Other: Scraping and straightening of the crown and root and rinsing with mouthwashes

INTERVENTIONS:
Other: Scraping and straightening of the crown and root and rinsing with mouthwashes — Patients will answer a questionnaire about their socioeconomic conditions, and soon after undergoing the examination for bleeding, probing, clinical attachment level, probing depth and plaque index for initial clinical evaluation. Basic periodontal treatment will be carried out with the same operator (blind to the treatments performed), with complete removal of plaque and calculi, prophylaxis with pumice and prophylactic paste and oral hygiene instructions. After basic periodontal treatment, patients will be randomly divided based on a draw with closed, opaque and non-translucent envelopes, into 3 groups according to the supporting treatments: G1 - patients who will receive mouthwashes with saline solution; G2 - patients who will be rinsed with 0.12% chlorhexidine and G3 - patients who will be treated with PHTALOX®.

SUMMARY:
Periodontitis is a chronic and destructive inflammation that leads to the loss of tissue supporting the teeth, the periodontium, and possibly tooth loss and edentulism. Its etiology is related to an overload on the host's defense mechanisms, consequent to the accumulation of plaque or suppression of the immune system. Standard treatment for periodontitis includes scaling and root planing (RAR) and possible association with therapeutic adjuvants such as systemic and local antimicrobials. However, the use of these drugs supporting the treatment of periodontitis, has shown adverse effects such as loss of taste, soft tissue burn, pain, xerostomia, supragingival calculus formation and change in staining of teeth, restorations, prostheses and tongue. Other effects not as common as mucosal ulcerations, desquamative lesions, urticaria, dyspnea, anaphylactic shock and swellings reversible effects in the parotid glands and lips have also been observed and reported in the literature. Thus, there is a need for new adjuvant therapies, which cause less effects side effects and that are more effective in the treatment of periodontitis and in the maintenance of oral health.

The commercial product PHTALOX® is a phthalocyanine dental mouthwash that has a spectrum of action based on the formation of reactive oxygen that acts by inhibiting odor-causing substances, on microorganisms and on the mechanisms of coagulation and healing. Your supporting action in periodontal treatment may have promising potential. Thus, the purpose of this study clinical trial will be testing a formulation containing PHTALOX® for disease prevention and control Periodontal (PD). 30 patients will be recruited who will undergo scaling and straightening coronaroradicular (RAR), and after basic periodontal treatment will be randomly divided into 3 groups according to the supporting treatment: G1 - patients who will receive mouthwashes with physiological solution; G2 - patients who will receive 0.12% chlorhexidine mouthwash; G3 - patients who will be treated with PHTALOX®. Clinical reassessments of patients will be carried out before the treatments, and at 15, 30 and 60 days after the performance of the RAR and beginning of the respective mouthwash. After data collection, intra and intergroup analyzes will be performed comparing the therapeutic results for the periodontal condition through the "Bioestat" program.

DETAILED DESCRIPTION:
PATIENT SELECTION

The research project will be submitted to the Ethics Committee for Research with Human Beings, at the Federal University of Alfenas (UNIFAL-MG), following the resolution of the National Health Council 466/2012.

Statistical planning was performed using the formula n = 1 + [2 * 10.51 * (0.2 / 0.172) ²], obtaining a number of approximately 30 patients, with a study power of 90%. This study will be clinical, double blind, involving patients aged between 18 and 50 years, who will be seen at the Periodontics Clinic of the Faculty of Dentistry, UNIFAL-MG and diagnosed with periodontitis. Secondary data will not be used for the study. After diagnosis, patients will read and sign the Informed Consent Form.

Patients will answer a questionnaire about their socioeconomic conditions, and soon after undergoing the examination for bleeding, probing, clinical attachment level, probing depth and plaque index for initial clinical evaluation. Basic periodontal treatment will be carried out with the same operator (blind to the treatments performed), with complete removal of plaque and calculi, prophylaxis with pumice and prophylactic paste and oral hygiene instructions. After basic periodontal treatment, patients will be randomly divided based on a draw with closed, opaque and non-translucent envelopes, into 3 groups according to the supporting treatments: G1 - patients who will receive mouthwashes with saline solution; G2 - patients who will be rinsed with 0.12% chlorhexidine and G3 - patients who will be treated with PHTALOX®. Each group will consist of the same number of patients, that is, 10. Patients will receive 140 mL of the substances, to be used for 7 days, twice a day.

Clinical reassessments of patients will be made before the treatments, and at 15, 30 and 60 after the performance of the RAR and beginning of the respective mouthwashes.

INSTRUCTIONS TO PATIENTS

Patients will be instructed on how they will use therapeutic adjuvants, according to the product to be used. In the act of orientation, the patient will use the adjunct for further explanation and standardization.

Treated patients will be instructed to use the product twice a day for 7 days, one in the morning and one in the evening, 30 minutes after brushing and flossing. The mouthwash should be carried out for 30 seconds with 10 mL of the solution corresponding to the group. All products must be completely expelled after rinsing. No product can be diluted in water and, after its use, the patient cannot eat or drink any liquid for at least 30 minutes. The patient will be advised that any signs of irritation, pain or other adverse effects that may appear are reported to the research group for evaluation.

As for oral hygiene habits, the patient should brush their teeth at least 3 times a day and floss at least once a day. The mean value of the frequency of oral hygiene habits will be collected at the end of the treatment, as well as information regarding gender, age, socioeconomic level, education level and number of teeth, for further analysis.

In addition, patients will be evaluated through the Community Periodontal Index, O' Leary Index and Bleeding Index on Probing.

STATISTICAL ANALYSIS

After collecting the primary data, intra and intergroup analyzes will be performed comparing socioeconomic results, periodontal condition, and treatments in isolation and their interrelationships through the "Bioestat" program.

ELIGIBILITY:
Exclusion criteria:

* Individuals who do not wish to complete the treatment protocol
* Individuals with healthy periodontium
* pregnant women
* Infants
* Individuals who use drugs
* Individuals with systemic alterations
* Individuals who used antibiotics in the last 3 months
* Individuals with systemic diseases that require antibiotic prophylaxis before periodontal therapy
* Immunosuppressed individuals

Inclusion criteria:

* Individuals of both sexes
* Individuals without a history of systemic complications for more than 6 months
* Individuals with no recent history of drug use
* Systemically healthy individuals
* Individuals with periodontal disease

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in COMMUNITY PERIODONTAL INDEX (CPI) | At Baseline ,15, 30 and 60 days after the performance of the RAR
  Will be obtained through periodontal probing in millimeters (mm) in six points of the index teeth. It allows evaluating the periodontal condition regarding health, bleeding and presence of calculus or pocket. The objective is to evaluate the improvement of periodontal conditions of patients.
Change in O' LEARY INDEX | At 15, 30 and 60 days after the performance of the RAR
  will be obtained by the percentage (%) of bacterial plaque on the faces of all teeth present in the oral cavity, dividing the number of surfaces containing plaque by the total number of surfaces evaluated. The objective is to evaluate the improvement of periodontal conditions of patients.
Change in PROBING BLEEDING INDEX (ISS) | At 15, 30 and 60 days
  Will be obtained by the percentage (%) of bleeding represented by the number of bleeding tooth surfaces, divided by the number of tooth surfaces examined. The objective is to evaluate the improvement of periodontal conditions of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Leandro Fernandes, Doctor, Principal Investigator — UNIFAL-MG
Locations (1):
- Unifal-Mg, Alfenas, Minas Gerias, Brazil

IPD SHARING:
Plan to Share IPD: No
At first, the data will not be shared with other researchers. This will take place at the time of publication of the research results.

REFERENCES:
- See also: Related Info — http://pubmed.ncbi.nlm.nih.gov/31941021/